CLINICAL TRIAL: NCT02496130
Title: A Partners Prospective Study Assessing the Perioperative Outcomes of Common Methods of Minimally Invasive Contained Tissue Extraction
Brief Title: Perioperative Outcomes of Common Methods of Minimally Invasive Contained Tissue Extraction
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jon I. Einarsson, Chief, Division of Minimally Invasive Gynecology, Brigham and Women's Hospital
Other Study IDs: 2015P000230
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Hysterectomy
Keywords: minilaparotomy; morcellation; laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- minilaparotomy: Subjects in this group will have tissue (uterus) extracted via mini-laparotomy incision with knife morcellation. Morcellation will be performed within a containment system. Method of extraction/group assignment will be determined clinically by the operating surgeon based on patient characteristics and patient preference.
- vaginal extraction: Subjects in this group will have tissue (uterus) extracted via vaginal extraction with knife morcellation. Morcellation will be performed within a containment system. Method of extraction/group assignment will be determined clinically by the operating surgeon based on patient characteristics and patient preference.

SUMMARY:
The goal of this study is to compare common methods of tissue extraction at the time of minimally invasive surgery.

DETAILED DESCRIPTION:
The goal of this study is to compare common methods of tissue extraction at the time of minimally invasive surgery, including vaginal extraction and mini-laparotomy; both performed within a containment system. The primary aim is to assess return to normal daily activities after each of the surgical techniques. Return to daily activities will be recorded on a post-operative patient activity diary recording the following tasks: a) work (if applicable), b) domestic tasks, c) driving a vehicle (if applicable) and d) physical exercise (if applicable). Additional information regarding post-operative pain (measured on a Likert scale), potential complications of each technique, such as tearing of the bag or leakage, and peri- and post-operative outcomes will be collected. In order to aid in detection of leakage, blue dye (either indigo carmine or methylene blue) will be added to the containment bag prior to morcellation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* eligible to undergo laparoscopic Hysterectomy, as determined clinically by the operating surgeon

Exclusion Criteria:

* suspected malignancy
* medical illness precluding laparoscopy
* inability to give informed consent
* allergy to indigo carmine or methylene blue dye

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 adult women scheduled to undergo a laparoscopic hysterectomy
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Return to daily activities | assessed between 2 and 6 weeks after surgery (at post-op visit)
  Return to daily activities will be recorded on a post-operative patient activity diary recording the following tasks: a) work (if applicable), b) domestic tasks, c) driving a vehicle (if applicable) and d) physical exercise (if applicable).

SECONDARY OUTCOMES:
OR Time | At the time of surgery
  minutes from procedure start to procedure end
Estimated Blood Loss | At the time of surgery
  ml of blood loss based on surgeon estimate
Spillage of the morcellated tissue or fluids in the abdomen and pelvis | At the time of surgery
  Following morcellation and removal of the bag, the abdomen and pelvis will be carefully examined for any signs of spillage of fluid, tissue or blue dye as well as the integrity of the containment system by the surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Jon I Einarsson, MD, PhD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT02496130/Prot_000.pdf